CLINICAL TRIAL: NCT03364634
Title: Intracranial Pressure After Decompressive Craniectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Alexander Lilja-Cyron, MD, PhD fellow, Rigshospitalet, Denmark
Other Study IDs: ICPinDCv1.1; H-15009654 (Other: The Regional Committee on Health Research Ethics)
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Traumatic Brain Injury; Middle Cerebral Artery Stroke; Intracranial Hemorrhages; Intracranial Hypertension
Keywords: decompressive craniectomy; intracranial pressure; icp; telemetry; telemetric
MeSH Terms: conditions — Brain Injuries, Traumatic; Infarction, Middle Cerebral Artery; Intracranial Hemorrhages; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intracranial pressure monitoring — Weekly ICP monitoring sessions beginning at discharge from the neuro-intensive care unit and carried out until 1 month after cranioplasty.

SUMMARY:
Observational study to investigate the natural course of intracranial pressure (ICP) after decompressive craniectomy (DC) using long-term telemetric ICP monitoring. Patients will have continuous ICP measurement performed during the admission to the neuro-intensive care unit (NICU) and after discharge weekly measurements sessions will be performed before and after cranioplasty.

DETAILED DESCRIPTION:
Several studies have investigated and documented the effect of DC in lowering ICP in intracranial hypertension following acute brain injuries, e.g. severe traumatic brain injury. But the natural course of ICP in these patients after the acute phase in the NICU has never been investigated. Clinical experience suggests that a DC affects cerebrospinal fluid circulation and ICP, e.g. causing hydrocephalus or subdural hygromas.

The aim of this observational study is to document the natural course of ICP following DC and to investigate the effect of cranioplasty on ICP. This is done by implantation of a telemetric ICP sensor and weekly follow-up monitoring sessions after discharge from the NICU until 1 month after cranioplasty. The monitoring sessions will include standardized body positions to investigate postural ICP changes before and after cranioplasty. The project will also provide experience with telemetric ICP monitoring during the acute phase in a NICU setting.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* scheduled for a decompressive hemicraniectomy for elevated ICP or signs of intracranial herniation

Exclusion Criteria:

* skin damage in the frontal area where the telemetric ICP sensor is implanted
* lack of informed consent from next-of-kin or the patient's general practitioner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for a decompressive hemicraniectomy for elevated ICP (e.g. following severe traumatic brain injury) or signs of intracranial herniation (e.g. following cerebral edema in patients with middle cerebral artery infarction).
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Intracranial pressure variations | Weekly monitoring sessions from discharge from the neuro-intensive care unit to 1 month after cranioplasty
  ICP is measured in standardized body positions to investigate postural changes after decompressive craniectomy and following cranioplasty

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website of Copenhagen CSF Study Group — http://www.cphcsf.dk
- See also: Website of Rigshospitalet (Copenhagen University Hospital), where the study is carried out — https://www.rigshospitalet.dk/english